CLINICAL TRIAL: NCT06037369
Title: The Effectiveness of a Short Message-based Customized Standardized Education Program in Promoting Wound Healing and Quality of Life of Patients With Diabetic Foot Ulcers
Brief Title: The Short Message-based Customized Standardized
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funds and the lack of significant results from the pilot test, we terminated the study.
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chin yenfan, assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRPD1N0241; NSTC112-2314-B-182-028 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: short message; wound healing; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): At each visit of the research subjects to plastic clinic, the research team record the attending prescriptions and patient educations given by the medical team members, and evaluate whether the research subjects and caregivers need additional mental support or not. Then, according to the above evaluation and records, items of a designed patient education menu will be selected, and the selected patient education messages will be sent according to the transmission frequency and time period proposed by the research object
  Interventions: Behavioral: customized standardized educational program sent by LINE software.
- comparison (No Intervention): Routine care

INTERVENTIONS:
Behavioral: customized standardized educational program sent by LINE software. — At each visit of the research subjects to plastic clinic, the research team record the attending prescriptions and patient educations given by the medical team members, and evaluate whether the research subjects and caregivers need additional mental support or not. Then, according to the above evaluation and records, items of a designed patient education menu will be selected, and the selected patient education messages will be sent according to the transmission frequency and time period proposed by the research object.
  Arms: intervention

SUMMARY:
The purpose of this study is to develop a short message-based customized standardized diabetic foot ulcer patient education program, and to test the effect of the program on diabetic foot ulcer self-management behavior, self-efficacy, wound prognosis, and quality of life.

A customized standardized patient education module will be developed, and then the effectiveness evaluation will be carried out. A randomized controlled study design will be adopted, and more than 30 outpatients with diabetic foot ulcers are expected to be recruited. The control group will receive routine care, while the experimental group will receive a short message-based customized standardized diabetic foot ulcer patient education program after their outpatient visits. Subjects will be followed up for eight weeks, and the Mann-Whitney U test and Fisher's correct probability test will be used to evaluate the effectiveness of the intervention.

DETAILED DESCRIPTION:
The diabetic foot ulcer need complex treatment, and is with poor prognosis, thus it consumes medical resources and impedes the quality of life of patients. Most of the time, patients are required to perform diabetic foot ulcer self-management at home. However, their self-management behaviors are inadequate.

Individualized patient education message can promote and maintain appropriate diabetes self-management behaviors of patients. The short message-based customized standardized patient education program combines several smartphone message-based standardized educational contents to construct a customized patient education program which is according to the needs of patients, thus providing individualized patient education in a timely manner. The short message-based customized standardized patient education program may improve the diabetic foot ulcers self-management behavior and the self-efficacy on diabetic foot ulcers self-management, thereby promoting wound healing and improving quality of life.

The purpose of this study is to develop a short message-based customized standardized diabetic foot ulcer patient education program, and to test the effect of the program on diabetic foot ulcer self-management behavior, self-efficacy, wound prognosis, and quality of life.

The innovation of this study are as follows：our intervention is the first program in the world that (1) provides timely and individualized patient education in a customized standardized way, and (2) provides short message-based patient education for prevention and treatment of diabetic foot ulcers.

A customized standardized patient education module will be developed, and then the effectiveness evaluation will be carried out. A randomized controlled study design will be adopted, and more than 30 outpatients with diabetic foot ulcers are expected to be recruited. The control group will receive routine care, while the experimental group will receive a short message-based customized standardized diabetic foot ulcer patient education program after their outpatient visits. Subjects will be followed up for eight weeks, and the Mann-Whitney U test and Fisher's correct probability test will be used to evaluate the effectiveness of the intervention.

ELIGIBILITY:
The inclusion criteria are:

* Outpatients with foot ulcers
* Diagnosed as diabetic patients
* Can be interviewed in Mandarin or Taiwanese.

The exclusion criteria are:

* It is expected that there is no need to return to the clinic at the eighth week after the baseline, or the number of return visits within eight weeks will be less than two times
* Patient and family members living with him/her do not use a smart phone
* Being unable to read text messages on mobile phone, or with impaired hearing, could not answer the phone
* Impaired fine hand movements, unable to click on mobile phone text messages
* Unwilling to use the communication software LINE to receive text messages.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yenfan Chin, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Comparison
Started | 16 | 15
Completed | 16 | 14
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.88 (9.80) | 60.0 (9.61) | 55.29 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 16 | 15 | 31
The wound area [Mean (Standard Deviation); unit: cm2] — Wound size is calculated by multiplying the length of the longest part of the wound by its vertical The longest width in the direction. For irregular-shaped areas, take pictures and use image statistics software to calculate the area.
  Wound meter measurements to assess subsequent changes
  cm2 | 4.5013 (6.49684) | 3.8820 (5.05084) | 4.4342 (5.69722)
Quality of life [Median (Inter-Quartile Range); unit: units on a scale] — Measuring quality of life with the Wound QoL-14. This is the pretest data
  units on a scale | 18.5 [14.0 to 22.75] | 21.0 [15.0 to 30.0] | 19.0 [14.0 to 25.0]

OUTCOME MEASURES:

1. Primary Outcome: Whether the Wound Shrinks
Description: In this study, Subtract the pre-measurement area from the post-measurement area to assess whether the wound has shrunk.
Time Frame: baseline and after four, eight weeks
Population: One participant was lost at four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
Participants
  wound shrinks at four weeks | 10 | 12
  wound shrink at eight weeks | 11 | 14

2. Primary Outcome: Diabetes-related Foot Ulcer Quality of Life
Description: Questionnaire on quality of life with chronic wounds (Wound QoL-14) will be used at four weeks and eight weeks after baseline to evaluate the change of QOL. Questionnaire on quality of life with chronic wound (Wound-QoL) has 14 items to measure the quality of life of patients with chronic wounds. Using the 5-point Likert scale, the patients were asked to report their chronic wounds in the past seven days, ranging from 0 (not at all) to 4 (very affected), with higher average scores indicating poorer quality of life. The range of scores is 0 to 56.
Time Frame: Baseline and after four, eight weeks
Population: One participants lost follow-up at four weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
score on a scale
  QoL at four weeks | 15.5 [13.0 to 22.25] | 16.5 [14.75 to 30.50]
  QoL at eight weeks | 12.50 [9.50 to 16.00] | 15.00 [10.50 to 28.25]

3. Secondary Outcome: Diabetes-related Foot Ulcer Self-management Behavior
Description: In this study, "Diabetes-related Foot Ulcer Self-Management Behavior Scale" (DFUSMB), will be used to measure DFU self-management behavior at four weeks and eight weeks after baseline.
  The DFUSMB measures behaviors that promote wound healing and prevent wound deterioration with 18 items in total, using the five-point Likert scale. "Never", "Seldom", "Sometimes", "Often" and "Always" are scored from 1 to 5 respectively. Reverse questions are scored in reverse, and the higher the total score, the better the self-management behavior of DFUs. In this study, we only collected the wound management subscale scores. The 7-item subscale score ranges 7-35. The DFUSMB has sufficient reliability and validity.
Time Frame: Baseline and after four, eight weeks
Population: One participant lost at four weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
score on a scale
  DFU self-management behavior at four weeks | 33 [31.00 to 34.00] | 34 [32.00 to 34.25]
  DFU self-management behavior at eight weeks | 34 [32.25 to 34.75] | 34 [31.50 to 35.00]

4. Secondary Outcome: Diabtes-related Foot Ulcer Self-management Self-efficacy
Description: We used 11 questions to measure the diabtes-related foot ulcer self-management self-efficacy, using an 11-point scale, with 0 indicating no confidence at all and 10 indicating complete confidence. Higher scores reflect higher self-efficacy. The sum score of the above 11 items indicates the DFU self-management self-efficacy with range from 0 to 110.
Time Frame: Baseline and after four, eight weeks
Population: One participant lost at four weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
score on a scale
  self-management self-efficacy at four weeks | 97.5 [93.625 to 103] | 95.0 [88.125 to 103.25]
  self-management self-efficacy at eight weeks | 98.5 [93.5 to 102.5] | 98.0 [87.0 to 102.25]

5. Secondary Outcome: Diabetes Self-care Behaviors
Description: The summary of diabetes self-care activity questionnaire (SDSCA) In this study, the summary of diabetes self-care activity questionnaire (SDSCA) will be used. The SDSCA questionnaire was developed by Deborah Toobert. It focuses on general diet, diabetes-specific diet, physical activity, blood-glucose testing, foot care, and smoking. The instrument assesses the absolute frequency or consistency of ten diabetes health-related regimen behaviors (e.g., number of days per week on which respondents engage in physical activity sessions; number of days in past 7 days respondents ate five or more servings of fruits and vegetables). Reverse questions are scored in reverse, and the higher the total score, the better the diabetes self-care activity. The total SDSCA score ranges 1-63.
Time Frame: Baseline and after four, eight weeks
Population: One participant lost at four weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
score on a scale
  SDSCA at four weeks | 37.0 [31.0 to 47.5] | 35.0 [26.75 to 42.25]
  SDSCA at eight weeks | 35.50 [30.0 to 49.75] | 35.0 [28.75 to 39.25]

6. Secondary Outcome: Diabetes-related Foot Self-care Behavior
Description: In this study, "Diabetic Foot Self-Care Behavior Scale" (DFSBS) will be used to measure diabetes-related foot self-care behavior at four weeks and eight weeks after baseline. The DFSBS has 7 questions, asking the participants how often they perform foot care behaviors. The total DFSBS score ranges 7-35. The higher the score, the better the foot care behavior. The DFSBS has sufficient reliability and validity.
Time Frame: Baseline and after four, eight weeks
Population: One participant lost at four weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 16 | 14
score on a scale
  Diabetes-related foot self-care behavior at four weeks | 22.0 [17.0 to 25.0] | 23.0 [17.25 to 25]
  Diabetes-related foot self-care behavior at eight weeks | 22.0 [19.5 to 25.0] | 22.50 [17.25 to 24.25]

ADVERSE EVENTS:
Time Frame: 4, 8 weeks
Description: The number of participants at risk for Serious Adverse Events is 31. The number of participants at risk for All-Cause Mortality is 31. The number of participants at risk for Other (Not Including Serious) Adverse Events is 31.
Arm/Group | Intervention | Comparison
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT06037369/Prot_SAP_000.pdf